CLINICAL TRIAL: NCT03312023
Title: A Phase II Open-Label Study of Ledipasvir/Sofosbuvir for 12 Weeks in Subjects With Hepatitis B Virus Infection
Brief Title: Ledipasvir/Sofosbuvir for Hepatitis B Virus Infection
Acronym: APOSTLE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Joel Chua, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00074723
Record Dates: First submitted 2017-09-29; First posted 2017-10-17 (Actual); Results first posted 2021-08-25 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-08

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; HBsAg; Ledipasvir/Sofosbuvir; Hepatitis B treatment
MeSH Terms: conditions — Hepatitis B | interventions — ledipasvir; Sofosbuvir; Tablets; ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Intervention Model Description: Open-label Study, multi-arm
Masking Description: Ten potential subjects for Groups C and D will be randomized in a 1:1 fashion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group A (LDV/SOF for low replicative HBV) (Experimental): 12 week treatment with ledipasvir/sofosbuvir (Harvoni) for chronic hepatitis B in low replicative state.
  Interventions: Drug: Ledipasvir 90 MG / Sofosbuvir 400 MG Oral Tablet [Harvoni]
- Group B (LDV/SOF for viral suppressed HBV) (Experimental): 12 week treatment with ledipasvir/sofosbuvir (Harvoni) for chronic hepatitis B, virally suppressed.
  Interventions: Drug: Ledipasvir 90 MG / Sofosbuvir 400 MG Oral Tablet [Harvoni]
- Group C (SOF for low replicative HBV) (Experimental): 12 weeks treatment with sofosbuvir (Sovaldi) for chronic hepatitis B in low replicative state.
  Randomized 1:1 with Group D.
  Interventions: Drug: Sofosbuvir 400 MG [Sovaldi]
- Group D (LDV for low replicative HBV) (Experimental): 12 weeks treatment with ledipasvir for chronic hepatitis B in low replicative state.
  Randomized 1:1 with Group C.
  Interventions: Drug: Ledipasvir 90 MG

INTERVENTIONS:
Drug: Ledipasvir 90 MG / Sofosbuvir 400 MG Oral Tablet [Harvoni] — 1 pill once daily for 12 weeks for Group A
  Other Names: Harvoni
  Arms: Group A (LDV/SOF for low replicative HBV); Group B (LDV/SOF for viral suppressed HBV)
Drug: Sofosbuvir 400 MG [Sovaldi] — 1 pill once daily for 12 weeks for Group C
  Other Names: GS-7977
  Arms: Group C (SOF for low replicative HBV)
Drug: Ledipasvir 90 MG — 1 pill once daily for 12 weeks for Group D
  Other Names: GS-5885
  Arms: Group D (LDV for low replicative HBV)

SUMMARY:
The goals of therapy against chronic hepatitis B are to decrease the morbidity and mortality related to chronic HBV infection. Currently available antiviral therapy can suppress viral replication but only a small proportion attain functional cure, which is defined as HBV surface antigen-to-antibody seroconversion. Hepatitis B surface antigen (HBsAg) is a marker of persistent hepatitis B infection.

It has been observed that patients who had both hepatitis B and hepatitis C, and who were treated for their hepatitis C with 12 weeks of ledipasvir/sofosbuvir for had a decline in HBsAg levels. This study hypothesizes that a similar decrease would be seen in mono-infected hepatitis B subjects over the course of 12 weeks treatment with ledipasvir/sofosbuvir.

ELIGIBILITY:
INCLUSION CRITERIA

Participants in Groups A, C & D (Chronic HBV, low replicative state not requiring treatment):

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18 or older at screening
4. Diagnosed with chronic hepatitis B infection defined as one of the following:

   1. HBsAg or HBV DNA positivity for at least 6 months
   2. Medical records indicating a chronic HBV infection
5. HBeAg negative at screening
6. HBV DNA > lower level of quantitation (LLOQ)
7. Quantitative HBsAg at least 10 IU/mL at screening
8. Ability to take oral medication and be willing to adhere to the twelve week study drug regimen
9. For females of reproductive potential: usual practice of complete abstinence from sexual intercourse with a member of the opposite sex OR use of at least one form of highly effective contraception for at least 1 month prior to enrollment and agreement to use such a method during study participation and for an additional 30 days after the end of study drug administration
10. For males of reproductive potential: usual practice of complete abstinence from sexual intercourse with a member of the opposite sex OR use of at least one form of highly effective contraception for at least 1 month prior to enrollment and agreement to use such a method during study participation and for an additional 14 days after the end of study drug administration
11. Ability to communicate effectively with the study investigator and key staff
12. Medical management provided by a primary care provider
13. Ability to store medications at a room temperature of less than 86 degrees Fahrenheit
14. Not on antiviral therapy or requiring treatment for HBV during screening

Participants in Group B (Chronic HBV, virally suppressed):

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18 or older at screening
4. Diagnosed with chronic hepatitis B infection defined as one of the following:

   1. HBsAg or HBV DNA positivity for at least 6 months
   2. Medical records indicating a chronic HBV infection
5. Receiving oral anti-HBV medications (either tenofovir alafenamide, tenofovir disoproxil fumarate, entecavir, or a combination of no more than 2 of these agents) for at least three months prior to enrollment
6. HBV DNA ˂ lower level of quantitation (LLOQ) at screening and for at least three months prior
7. Quantitative HBsAg at least 10 IU/mL at screening
8. Ability to take oral medication and be willing to adhere to the twelve week study drug regimen
9. For females of reproductive potential: usual practice of complete abstinence from sexual intercourse with a member of the opposite sex OR use of at least one form of highly effective contraception for at least 1 month prior to enrollment and agreement to use such a method during study participation and for an additional 30 days after the end of study drug administration
10. For males of reproductive potential: usual practice of complete abstinence from sexual intercourse with a member of the opposite sex OR use of at least one form of highly effective contraception for at least 1 month prior to enrollment and agreement to use such a method during study participation and for an additional 14 days after the end of study drug administration
11. Ability to communicate effectively with the study investigator and key staff
12. Medical management provided by a primary care provider
13. Ability to store medications at a room temperature of less than 86 degrees Fahrenheit

EXCLUSION CRITERIA

1. Coinfection with hepatitis C, hepatitis D or human immunodeficiency virus (HIV)
2. Pregnancy or lactation
3. Known allergic reactions to sofosbuvir or ledipasvir
4. Treatment with another investigational drug or other intervention within three months
5. Evidence of cirrhosis or hepatic decompensation such as:

   * Platelets less than 100,000 /mm3
   * Albumin less than 3.5 g/dL
   * INR greater than 1.7 or Prothrombin time of 1.5 times the upper limit of normal (ULN)
   * Total bilirubin of 1.5 times the upper limit of normal
   * FibroTest (or FibroSure®) of 0.75 or greater
6. Abnormal hematological and biochemical parameters at screening including:

   * White blood cell count less than 2500 cells/uL
   * Absolute neutrophil count (ANC) less than 1,000 cells/mm3 (less than 750 mm3 for African or African-American subjects)
   * Hemoglobin less than 12 g/dL for males, less than 11 g/dL for females
   * AST or ALT of two times the upper limit of normal
   * Estimated GFR less than 50 mL/min
   * Glycosylated hemoglobin (HbA1c) greater than 8.5%
7. Current or prior history of any of the following:

   * Immunodeficiency disorders or autoimmune disease (e.g. Systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel diseases, sarcoidosis, psoriasis of greater than mild severity)
   * Severe pulmonary disorders, significant cardiac diseases
   * Gastrointestinal disorder with post-operative condition that could interfere with the absorption of the study drugs
   * Significant psychiatric illness that in the judgment of the Investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent
   * Any malignancy diagnosed within 5 years (not including recent localized treatment of squamous or non-invasive basal cell skin cancer; cervical carcinoma in situ appropriately treated prior to screening)
   * Solid organ transplantation
   * Poor venous access
8. Screening ECG with clinically significant findings
9. Evidence of HCC (e.g., α fetoprotein > 50ng/mL or radiologic evidence)
10. Clinically significant illicit drug or alcohol abuse within 12 months of screening. Subjects on methadone maintenance treatment or prescribed opioid may be included.
11. Use of amiodarone within 90 days of enrollment; or carbamazepine, phenytoin, phenobarbital, oxcarbazepine, rifabutin, rifampin, rifapentine, St. John's wort, rosuvastatin, or interferon within 30 days of enrollment or expected use of these prohibited drugs during study participation. Use of or expected need of proton-pump inhibitors more than 20 mg omeprazole equivalent or H2 receptor antagonist more than 40 mg famotidine BID equivalent within 7 days of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel V Chua, MD, Principal Investigator — University of Maryland, College Park
Locations (1):
- Institute of Human Virology (IHV), University of Maryland Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Group C (SOF for Low Replicative HBV): 12 weeks treatment with sofosbuvir (Sovaldi) for chronic hepatitis B in low replicative state.
  Randomized 1:1 with Group D.
  Sofosbuvir 400 MG [Sovaldi]: 1 pill once daily for 12 weeks for Group C
- Group D (LDV for Low Replicative HBV): 12 weeks treatment with ledipasvir for chronic hepatitis B in low replicative state.
  Randomized 1:1 with Group C.
  Ledipasvir 90 MG: 1 pill once daily for 12 weeks for Group D
Period: Overall Study
Arm/Group | Group A (LDV/SOF for Low Replicative HBV) | Group B (LDV/SOF for Viral Suppressed HBV) | Group C (SOF for Low Replicative HBV) | Group D (LDV for Low Replicative HBV)
Started | 8 | 5 | 4 | 4
Completed Week 12 ((end of treatment)) | 8 | 5 | 4 | 4
Completed | 8 | 5 | 4 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (LDV/SOF for Low Replicative HBV) | Group B (LDV/SOF for Viral Suppressed HBV) | Group C (SOF for Low Replicative HBV) | Group D (LDV for Low Replicative HBV) | Total
Number analyzed (Participants) | 8 | 5 | 4 | 4 | 21
Age, Continuous [Mean (Full Range); unit: years] | 47.3 [30 to 73] | 57.6 [42 to 73] | 43.5 [38 to 57] | 52.3 [42 to 61] | 50.0 [30 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 0 | 5
  Male | 7 | 3 | 2 | 4 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 5 | 4 | 4 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 3 | 0 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 2 | 3 | 3 | 12
  White | 1 | 0 | 1 | 1 | 3
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 5 | 4 | 4 | 21
Negative eAg [Count of Participants; unit: Participants] | 8 | 5 | 4 | 4 | 21
Normal ALT [Count of Participants; unit: Participants] | 8 | 5 | 3 | 4 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change of Serum Hepatitis B Surface Antigen (HBsAg as Measured in log10 IU/mL) Level as an Indicator of Antiviral Activity of Ledipasvir and/or Sofosbuvir in Subjects With Chronic Hepatitis B From Baseline to End of 12 Weeks Treatment.
Description: Subjects with chronic hepatitis B will be give 12 weeks of ledipasvir and/or sofosbuvir and their HBsAg will be measured at baseline, on each visits during therapy, and at end of therapy (week 12). The change (decline) in HBsAg from baseline to end of the 12 week treatment will be compared.
Time Frame: 12 weeks
Population: Intention to treat population - all subjects who have received at least one study drug.
Measure: Mean (Standard Deviation); unit: Log10 IU/mL
Arm/Group | Group A (LDV/SOF for Low Replicative HBV) | Group B (LDV/SOF for Viral Suppressed HBV) | Group C (SOF for Low Replicative HBV) | Group D (LDV for Low Replicative HBV)
Number analyzed (Participants) | 8 | 5 | 4 | 4
Log10 IU/mL | 0.39 (0.2) | 0.40 (0.3) | 0.19 (0.3) | -0.05 (0.1)

2. Primary Outcome: Incidence of Adverse Events Leading to Permanent Discontinuation of Ledipasvir and/or Sofosbuvir Treatment in Subjects With Chronic Hepatitis B Infection.
Description: Number of subjects who discontinued study drug due to adverse event
Time Frame: 12 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (LDV/SOF for Low Replicative HBV) | Group B (LDV/SOF for Viral Suppressed HBV) | Group C (SOF for Low Replicative HBV) | Group D (LDV for Low Replicative HBV)
Number analyzed (Participants) | 8 | 5 | 4 | 4
Participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Changes in Serum Hepatitis B Virus DNA Levels (HBV DNA as Measured in IU/mL) With Treatment of Ledipasvir and/or Sofosbuvir From Baseline to End of 12 Weeks of Treatment in Subjects With Chronic Hepatitis B Infection.
Description: Subjects with chronic hepatitis B will be give 12 weeks of ledipasvir and/or sofosbuvir and their serum hepatitis B DNA levels (HBV DNA) will be measured at baseline, on each visits during therapy, and at end of therapy (week 12). The change in HBV DNA levels from baseline to end of the 12 week treatment will be compared.
  Note: Group B (virally suppressed HBV subjects) - all had HBV DNA below the limit of detection; Hence, mean change was 0.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Log10 IU/mL
Groups:
- Group B (LDV/SOF for Virally Suppressed HBV): 12 weeks of treatment with ledipasvir/sofosbuvir (Harvoni) for chronical hepatitis B virally suppressed on HBV meds
Arm/Group | Group A (LDV/SOF for Low Replicative HBV) | Group B (LDV/SOF for Virally Suppressed HBV) | Group C (SOF for Low Replicative HBV) | Group D (LDV for Low Replicative HBV)
Number analyzed (Participants) | 8 | 5 | 4 | 4
Log10 IU/mL | 0.51 (0.6) | 0 (0) | 0.68 (0.4) | 0.21 (0.8)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Group A (LDV/SOF for Low Replicative HBV) | Group B (LDV/SOF for Viral Suppressed HBV) | Group C (SOF for Low Replicative HBV) | Group D (LDV for Low Replicative HBV)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/5 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/5 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 7/8 | 2/5 | 4/4 | 1/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (LDV/SOF for Low Replicative HBV) (N=8) | Group B (LDV/SOF for Viral Suppressed HBV) (N=5) | Group C (SOF for Low Replicative HBV) (N=4) | Group D (LDV for Low Replicative HBV) (N=4)
Headache (Nervous system disorders) | 4 (10) | 2 (3) | 1 (1) | 0 (0)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (3) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 1 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (5) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash, maculopapular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis, allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema, peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle strain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-18): https://cdn.clinicaltrials.gov/large-docs/23/NCT03312023/Prot_SAP_000.pdf